CLINICAL TRIAL: NCT06812559
Title: Progesterone Primed Ovarian Stimulation Versus Gonadotrophin-Releasing Hormone Antagonist in Women With Polycystic Ovarian Syndrome
Brief Title: Progesterone Primed Ovarian Stimulation Versus GnRH Antagonist Protocols in Women With Polycystic Ovarian Syndrome
Status: Completed | Type: Observational
Sponsor: El Shatby University Hospital for Obstetrics and Gynecology (Other)
Responsible Party: Principal Investigator, Aly Hussein, Principle investigator, El Shatby University Hospital for Obstetrics and Gynecology
Other Study IDs: PPOS vs Antagonist Protocols
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Controlled Ovarian Hyperstimulation; Polycystic Ovarian Syndrome
Keywords: PPOS versus antagonist protocol in PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Progesterone; Dydrogesterone; cetrorelix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Progesterone-primed ovarian stimulation Group: • A daily dose of 20 mg dydrogesterone (2 Duphastone 10 mg tablets) will be added from day 1 or 2 of the menstrual cycle and will be continued till the day of the GnRH agonist trigger.
  Interventions: Drug: Progesterone
- Antagonist protocol: • GnRH antagonist (Cetrotide 0.25 mg) subcutaneous injection will be added daily from the 6th day of ovarian stimulation and will be continued till the day of the GnRH agonist trigger.
  Interventions: Drug: GnRH antagonist (Cetrorelix)

INTERVENTIONS:
Drug: Progesterone — compare the use of the progesterone-primed ovarian stimulation protocol versus GnRH antagonist protocol in women with polycystic ovarian syndrome (PCOS) regarding the number of oocytes retrieved, percentage of MII oocytes, and the rate of good quality blastocysts available for cryopreservation.
  Other Names: Duphaston 10mg Tablets
  Groups: Progesterone-primed ovarian stimulation Group
Drug: GnRH antagonist (Cetrorelix) — Subcutaneous injection
  Other Names: Cetrotide 0.25mg
  Groups: Antagonist protocol

SUMMARY:
The purpose of this study is to compare the use of the progesterone-primed ovarian stimulation protocol versus GnRH antagonist protocol in women with polycystic ovarian syndrome (PCOS) regarding the number of oocytes retrieved, percentage of MII oocytes, and the rate of good quality blastocysts available for cryopreservation.

DETAILED DESCRIPTION:
The syndrome of polycystic ovary (PCOS) is a common endocrine disease. It accounts for about 80% of women with anovulatory infertility. In vitro fertilization (IVF) is a commonly used infertility treatment for PCOS patients who fail to conceive with ovulation induction or if there are concomitant infertility factors such as tubal damage or male subfertility.

Patients with polycystic ovary syndrome (PCOS) are at high risk of ovarian hyperstimulation syndrome (OHSS) during in vitro fertilization (IVF) / intracytoplasmic sperm injection (ICSI) treatment which may lead to cycle cancellation to prevent their high morbidity or death rates. Increasing evidence has confirmed that frozen embryo transfer (FET) is related to a lower risk of OHSS. The 'freeze-all' strategy is recommended for PCOS patients to reduce the potential of moderate/severe OHSS.

Controlled ovarian stimulation (COS) is a key step in assisted reproductive technology (ART). In addition to the use of gonadotropins to recruit multiple follicles, it is mandatory to use a drug to prevent luteinizing hormone (LH) surge and premature ovulation.

Early LH surge is a main cause of cycle cancellation during controlled ovarian stimulation (COH) for women receiving IVF/ICSI therapy. The release of LH causes ovulation in response to rapidly increasing levels of E2 in the normal cycle, and a premature LH increase may impair IVF/ICSI egg production.

Gonadotropin-releasing hormone (GnRH) antagonist protocol has emerged as a routine ovulation stimulation protocol in recent decades due to its comparable convenience, safety, and efficacy compared to GnRH agonists. GnRH antagonist protocol is now the most commonly used COS protocol in PCOS patients due to the significantly reduced risk of OHSS especially when gonadotropin-releasing hormone agonist (GnRHa) was used for ovulation trigger. The GnRH antagonists were used primarily to reduce the incidence of the early LH surge. However, GnRH antagonists are expensive and sometimes difficult to manage with high rates of cycle cancellation and premature LH surges.

In past decades, when IVF relied on fresh embryo transfer, progesterone could not be considered during COS as early exposure to progesterone could lead to embryo-endometrium asynchrony. Advances in vitrification have made cryopreservation and thawing of embryos in a reliable manner, which has eliminated concerns about the deleterious effects of progesterone exposure on endometrial receptivity. Although controversies remain regarding the selection of when to choose FET, the ''freeze-all'' strategy could make the use of P formulations for the suppression of premature LH surge during COH feasible regardless of the effects of P on endometrial receptivity. Therefore, the PPOS protocol may be a suitable option when fresh embryo transfer is not required.

Progesterone-primed ovarian stimulation is a recent stimulation protocol, which was first suggested in 2015 by Dr. Yanping Kuang of China, it is a novel ovarian stimulation system utilizing progestin coupled with exogenous gonadotrophin, and ovulation triggered by a GnRH agonist, via 'freeze-all' methods. Oral progestin are used as an alternative to GnRH antagonist to prevent premature LH surges during ovarian stimulation. This novel ovarian stimulation regimen has shown successful prevention of a premature LH surge in cycles followed by embryo cryopreservation. In addition, oral progestin has the advantage of being convenient, given orally, cheap, and available readily.

The mechanism of LH suppression using GnRH-ant or progestin is distinct. GnRH-ant administration could lead to rapid suppression of pituitary LH secretion by competitively blocking the GnRH receptor, with an obvious dose-dependent suppression effect. In contrast, the inhibition of LH levels with progestin is indirect by regulating the hypothalamus GnRH secretion and requires sufficient duration before estrogen priming.

ELIGIBILITY:
Inclusion Criteria:

1. Female age <37 years.
2. Body mass index (BMI) between (≥18 kg/m2 and ≤35 kg/m2).
3. Polycystic ovarian syndrome patients (according to Rotterdam criteria).
4. Patients suffering from primary or secondary infertility who are candidates for ICSI.

Exclusion Criteria:

1. Uncorrected Uterine factor of infertility: intrauterine adhesions, submucosal fibroids, and septate uterus.
2. Severe male factor infertility

Max Age: 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Female aged less than 37 years old, with PCOS and infertility
Study Population: History taking and examination:
  * Basal ultrasound scanning includes 3D assessment of the uterine cavity and a basal hormonal profile.
  * Semen analysis.
  Ovarian stimulation:
  * Will be on day 2 or 3 of the menstrual cycle
  * Using rFSH SC injections with a dose of 150 to 225 IU per day and highly purified hMG with a dose of 75 IU per day.
  These patients will be divided into two equal groups:
  Group 1 (Fixed GnRH antagonist protocol) (n= 50):
  • GnRH antagonist (Cetrotide 0.25 mg) SC injection will be added daily from the 6th day of COH and will be continued till the day of the GnRH agonist trigger.
  Group 2 (Progesterone-primed ovarian stimulation) (n= 50):
  • A daily dose of 20 mg dydrogesterone (2 Duphastone 10 mg tablets) will be added from day 1 or 2 of the menstrual cycle till day of trigger
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Number of oocytes retrieved (ovarian response). | Baseline
  Total number of oocytes retrieved (in both groups)
Percentage of MII oocytes. | Baseline
  Number of MII oocytes to the total number of oocytes retrieved (in both groups)
Rate of good-quality blastocysts available for cryopreservation | Baseline
  percentage of the number of good-quality blastocysts to the number of 2PN fertilized oocytes cultured

SECONDARY OUTCOMES:
Fertilization rate | Baseline
  Percentage of the number of MII oocytes microinjected which transform into 2PN
Rate of blastocyst formation | Baseline
  percentage of the number of blastocysts formed to the number of 2PN fertilized oocytes cultured
Clinical pregnancy rate after 1st FET | Baseline
  defined as elevated serum β-HCG (+) the presence of gestational sac(s) or fetal heartbeats (fetal pole) by ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Ismail E Khalifa, Ass.lecturer, Principal Investigator — Elshatby University hospital; Sherif S Gafaar, Professor, Principal Investigator — Elshatby University hospital
Locations (1):
- ELShatby University Hospital, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lainas TG, Sfontouris IA, Zorzovilis IZ, Petsas GK, Lainas GT, Alexopoulou E, Kolibianakis EM. Flexible GnRH antagonist protocol versus GnRH agonist long protocol in patients with polycystic ovary syndrome treated for IVF: a prospective randomised controlled trial (RCT). Hum Reprod. 2010 Mar;25(3):683-9. doi: 10.1093/humrep/dep436. Epub 2009 Dec 15. PMID 20008886
- [Background] Griesinger G, Diedrich K, Tarlatzis BC, Kolibianakis EM. GnRH-antagonists in ovarian stimulation for IVF in patients with poor response to gonadotrophins, polycystic ovary syndrome, and risk of ovarian hyperstimulation: a meta-analysis. Reprod Biomed Online. 2006 Nov;13(5):628-38. doi: 10.1016/s1472-6483(10)60652-9. PMID 17169171
- [Background] Al-Inany HG, Youssef MA, Ayeleke RO, Brown J, Lam WS, Broekmans FJ. Gonadotrophin-releasing hormone antagonists for assisted reproductive technology. Cochrane Database Syst Rev. 2016 Apr 29;4(4):CD001750. doi: 10.1002/14651858.CD001750.pub4. PMID 27126581
- [Background] Toftager M, Bogstad J, Lossl K, Praetorius L, Zedeler A, Bryndorf T, Nilas L, Pinborg A. Cumulative live birth rates after one ART cycle including all subsequent frozen-thaw cycles in 1050 women: secondary outcome of an RCT comparing GnRH-antagonist and GnRH-agonist protocols. Hum Reprod. 2017 Mar 1;32(3):556-567. doi: 10.1093/humrep/dew358. PMID 28130435
- [Background] Depalo R, Jayakrishan K, Garruti G, Totaro I, Panzarino M, Giorgino F, Selvaggi LE. GnRH agonist versus GnRH antagonist in in vitro fertilization and embryo transfer (IVF/ET). Reprod Biol Endocrinol. 2012 Apr 13;10:26. doi: 10.1186/1477-7827-10-26. PMID 22500852
- [Background] Messinis IE. Ovarian feedback, mechanism of action and possible clinical implications. Hum Reprod Update. 2006 Sep-Oct;12(5):557-71. doi: 10.1093/humupd/dml020. Epub 2006 May 3. PMID 16672246
- [Background] Zhou R, Dong M, Huang L, Wang S, Fan L, Liang X, Zhang X, Liu F. Comparison of cumulative live birth rates between progestin-primed ovarian stimulation protocol and gonadotropin-releasing hormone antagonist protocol in different populations. Front Endocrinol (Lausanne). 2023 Apr 18;14:1117513. doi: 10.3389/fendo.2023.1117513. eCollection 2023. PMID 37143731
- [Background] Pirtea P, de Ziegler D, Poulain M, Ayoubi JM. New Twists in Ovarian Stimulation and Their Practical Implications. Front Med (Lausanne). 2019 Sep 4;6:197. doi: 10.3389/fmed.2019.00197. eCollection 2019. PMID 31555650
- [Background] Zhu X, Ye H, Ye J, Fu Y. Progesterone protocol versus gonadotropin-releasing hormone antagonist protocol in women with polycystic ovarian syndrome undergoing in vitro fertilization treatments with frozen-thawed embryo transfer: a prospective randomized controlled trial. Ann Transl Med. 2021 Mar;9(5):387. doi: 10.21037/atm-20-1592. PMID 33842608
- [Background] Chen ZJ, Shi Y, Sun Y, Zhang B, Liang X, Cao Y, Yang J, Liu J, Wei D, Weng N, Tian L, Hao C, Yang D, Zhou F, Shi J, Xu Y, Li J, Yan J, Qin Y, Zhao H, Zhang H, Legro RS. Fresh versus Frozen Embryos for Infertility in the Polycystic Ovary Syndrome. N Engl J Med. 2016 Aug 11;375(6):523-33. doi: 10.1056/NEJMoa1513873. PMID 27509101
- [Background] Delvigne A, Rozenberg S. Epidemiology and prevention of ovarian hyperstimulation syndrome (OHSS): a review. Hum Reprod Update. 2002 Nov-Dec;8(6):559-77. doi: 10.1093/humupd/8.6.559. PMID 12498425
- [Background] Sultan C, Paris F. Clinical expression of polycystic ovary syndrome in adolescent girls. Fertil Steril. 2006 Jul;86 Suppl 1:S6. doi: 10.1016/j.fertnstert.2006.04.015. PMID 16798287
- [Background] Thessaloniki ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group. Consensus on infertility treatment related to polycystic ovary syndrome. Hum Reprod. 2008 Mar;23(3):462-77. doi: 10.1093/humrep/dem426. PMID 18308833
- [Background] Zhu X, Ye H, Fu Y. The Utrogestan and hMG protocol in patients with polycystic ovarian syndrome undergoing controlled ovarian hyperstimulation during IVF/ICSI treatments. Medicine (Baltimore). 2016 Jul;95(28):e4193. doi: 10.1097/MD.0000000000004193. PMID 27428219